CLINICAL TRIAL: NCT04901533
Title: Effect of Occipito-atlas-axis Manipulation on Oculomotricity in Individuals With Exophories
Brief Title: Cervical Manipulation (OAA Technique) in Exophories
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Lourdes Mª Fernández Seguín, Assistant Professor. Physiotherapy Department, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EXOFORIAS
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Exophoria
Keywords: cervical manipulation; disorder ocular motility; musculoeskeletal; strabismus
MeSH Terms: conditions — Exotropia; Ocular Motility Disorders; Strabismus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cervical manipulation (Experimental): The objective of this technique is to restore joint mobility between the joints of the occipital, first (atlas) and second cervical vertebra (axis). It is a technique performed in rotation on a vertical axis that passes through the odontoid process of the axis, without placing flexion or extension, and with very slight sidebending; it is done bilaterally.
  Interventions: Procedure: O-A-A
- Cranial Listening (Active Comparator): Cranial palpation maneuver
  Interventions: Procedure: cranial listening

INTERVENTIONS:
Procedure: O-A-A — patient is supine, and the therapist stands on the side to be manipulated. The cranial hand of the therapist globally grasps the patient's skull and turns the patient's neck on that same side. The caudal hand is placed on the patient's face. The technique is performed by an impulse in pure rotation on the side that the cervical region is rotated, with a helical movement.
  Arms: cervical manipulation
Procedure: cranial listening — The patient is in the supine position, and the therapist sitting at the head of the patient. The therapist places his hands on the head of the patient, the thumbs touch each other, without touching the vault cranial. A perception of the cranial rhythm is carried out passively.
  Arms: Cranial Listening

SUMMARY:
Objetive: to assess the efficacy of the occipito-atlas-axis cervical manipulation technique to correct ocular divergence in subjects with exophoria.

Design: quantitative, experimental, longitudinal and prospective study.

Subjects: subjects over 18 years of age, with exophorias, without heterotropies and who do not present a contraindication to cervical manipulation.

Methods:Subjects with this ocular mobility dysfunction are going to be evaluated objectively with the Alternate Cover Test. The ocular deviation will be measured at 40 cm and at 4 meters. The individuals who were part of the experimental group underwent the OAA manipulation technique, and to those who were part of the control group a placebo maneuver. Two measurements were taken from this moment, one immediately after the execution of the technique and another one week later.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of exophoria
* Being 18 years old.

Exclusion Criteria:

* Having heterotropia or have been treated for it.
* Present contraindication to manipulation (recent fractures, sprains, or dislocations, local tumor, rheumatic polyarthritis, Down syndrome, vertebrobasilar insufficiency, basilar impression, refusal to be manipulated).
* Having cervical manipulation before two weeks.

Ages: 18 Years to 57 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
exophoria with cover test at 40 cm | Changes from baseline to moment after intervention
  The exophoria will be evaluated in prismatic diopter.
  Using the cover alternate test, therapist will measure with a prism ruler the diopters that the subject requires to balance eye movement and that the eye does not move from the outside to the inside when looking at an object at 40 cm.
exophoria with cover test al 4 m | Changes from baseline to moment after intervention
  The exophoria will be evaluated in prismatic diopter. Using the cover alternate test, therapist will measure with a prism ruler the diopters that the subject requires to balance eye movement and that the eye does not move from the outside to the inside when looking at an object at 4 meters.

SECONDARY OUTCOMES:
exophoria with cover test at 40 cm (2) | Changes from baseline to 1 week after intervention
  The exophoria will be evaluated in prismatic diopter. Using the cover alternate test, therapist will measure with a prism ruler the diopters that the subject requires to balance eye movement and that the eye does not move from the outside to the inside when looking at an object at 40 cm.
exophoria with cover test al 4 m (2) | Changes from baseline to 1 week after intervention
  The exophoria will be evaluated in prismatic diopter. Using the cover alternate test, therapist will measure with a prism ruler the diopters that the subject requires to balance eye movement and that the eye does not move from the outside to the inside when looking at an object at 4 meters.

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes M Fernández-Seguín, PhD, Principal Investigator — University of Seville
Locations (1):
- Lourdes M Fernández-Seguín, Seville, Spain

REFERENCES:
- [Derived] Fernandez-Seguin LM, Peinado-Asensio M, Diaz-Mancha JA, Cortes-Vega MD, Heredia-Rizo AM. Short-Term Effect of Spinal Manipulation on the Magnitude of Exophoria in Adults Who Are Asymptomatic: A Randomized Controlled Trial. Phys Ther. 2023 Aug 1;103(8):pzad069. doi: 10.1093/ptj/pzad069. PMID 37347984